CLINICAL TRIAL: NCT06395701
Title: Retrospective Study Protocol on Bladder Cancer With Bladder Preservation Intent
Brief Title: Trimodality Treatment in Bladder Cancer
Status: Completed | Type: Observational
Sponsor: Consorci Sanitari de Terrassa (Other)
Responsible Party: Principal Investigator, Nicolas Feltes, M.D, Consorci Sanitari de Terrassa
Other Study IDs: TRIMODAL-VEJIGA
Record Dates: First submitted 2024-04-29; First posted 2024-05-02 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Bladder Cancer; Urinary Bladder Neoplasms; Bladder Disease
MeSH Terms: conditions — Urinary Bladder Neoplasms; Urinary Bladder Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Radiation: radioteraphy and chemotherapy after RTU --trimodality therapy-- — TMT ( trimodality treatment) consists of complete and maximal TURBT of the bladder tumor, followed by definitive radiotherapy combined with a radiosensitizing agent.

SUMMARY:
Bladder cancer is a malignant disease that affects a large number of people worldwide. An increase in the incidence of this type of cancer has been observed in recent decades, leading to a growing interest in understanding its risk factors, clinical evolution, and possible treatment approaches. This retrospective study aims to retrospectively analyze a cohort of patients diagnosed with muscle-invasive bladder cancer, in whom, after presentation at multidisciplinary oncology committees, the goal of curing the oncological disease while preserving the bladder is considered.

Trimodal therapy (TMT) is the most studied bladder preservation strategy, with oncological outcomes superior to those of isolated therapies (or monotherapies) such as transurethral resection of the bladder tumor (TURBT), radiotherapy, or chemotherapy. TMT consists of complete and maximal TURBT of the bladder tumor, followed by definitive radiotherapy combined with a radiosensitizing agent.

Objectives The main objective is to retrospectively analyze the effectiveness and safety of the trimodal approach in our setting. Collecting and analyzing data from patients treated in our service will provide valuable insight into clinical outcomes and treatment tolerability in this context.

Materials and Methods

* Study Design A retrospective study will be conducted using data from medical records of patients diagnosed with bladder cancer from 2014 to 2022 and treated with radiotherapy in our Radiation Oncology Service. Demographic data, medical history, risk factors, clinical characteristics, treatments received, and clinical outcomes will be collected.
* Study Population The study population will include all patients with confirmed diagnoses of non-metastatic muscle-invasive bladder cancer.

DETAILED DESCRIPTION:
• Inclusion Criteria Adult patients (over 18 years old) with histologically confirmed diagnosis of bladder cancer.

Criteria for selecting optimal candidates for trimodal therapy-assessment in Uro-Oncology committees.

-Functional and compatible bladder at the start of the study.

Criteria related to the tumor:

* cT2
* Unifocal tumor with a maximum diameter < 7 cm.
* Single tumor.
* Absence of extensive associated carcinoma in situ (CIS).
* Absence of bilateral hydronephrosis.
* Absence of lymphovascular invasion.
* Attempt at macroscopically complete TURBT of the bladder (incomplete does not exclude bladder preservation).

Availability of complete medical records, including demographic data, medical history, imaging study results, treatment details, and follow-up.

* Data Collection Data will be retrospectively collected from patients' electronic medical records. Standardized forms will be used to record relevant data, including demographic information, medical history, imaging study results, treatment details, and follow-up.
* Statistical Analysis Descriptive analysis of the data will be performed to summarize the characteristics of the study population and clinical outcomes. Appropriate statistical tests will be used to compare patient subgroups and assess the association between variables of interest and clinical outcomes.
* Ethical Considerations This study will be conducted following the ethical principles established in the Helsinki Declaration. Approval will be obtained from our hospital's Ethics Committee.
* Study Limitations Potential limitations of this study may include inherent bias in retrospective studies, incomplete data in some medical records, and variability in treatments administered over time.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (over 18 years old) with histologically confirmed diagnosis of bladder cancer.

Criteria for selecting optimal candidates for trimodal therapy-assessment in Uro-Oncology committees.

-Functional and compatible bladder at the start of the study.

Criteria related to the tumor:

* cT2
* Unifocal tumor with a maximum diameter < 7 cm.
* Single tumor.
* Absence of extensive associated carcinoma in situ (CIS).
* Absence of bilateral hydronephrosis.
* Absence of lymphovascular invasion.
* Attempt at macroscopically complete TURBT of the bladder (incomplete does not exclude bladder preservation).

Availability of complete medical records, including demographic data, medical history, imaging study results, treatment details, and follow-up.

Exclusion Criteria:

* Not availability of complete medical records, including demographic data, medical history, imaging study results, treatment details, and follow-up.

Ages: 18 Years to 100 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with bladder cancer from 2014 to 2022 and treated with radiotherapy in our Radiation Oncology Service. Demographic data, medical history, risk factors, clinical characteristics, treatments received, and clinical outcomes will be collected
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2014-04-01 (Actual); Primary Completion 2024-06-02 (Actual); Study Completion 2024-06-02 (Actual)

PRIMARY OUTCOMES:
Local Control | 5-10 years
  Local Control assessed by RECIST criteria with TC, MRI or PET-scan

SECONDARY OUTCOMES:
Overall Survival | Overall Survival [ Time Frame: Participants should be followed continuously during 5-10 years Defined as the time from diagnose to the date of death from any cause.
  Defined as the time from diagnose to the date of death from any cause.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital de Terrassa, Terrassa, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No